CLINICAL TRIAL: NCT03143582
Title: Examining the Effects of a Team-based Running Program on the Mental Health and Cognition of Emerging Adults: A Pilot Study
Brief Title: Examining the Effects of a Team-based Running Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Juliana Tobon, Psychologist, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2785
Record Dates: First submitted 2017-04-28; First posted 2017-05-08 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Memory; Learning; Mood; Attention; Stress; Sleep
MeSH Terms: interventions — Running; Exercise

STUDY DESIGN:
Intervention Model Description: This is an open-label pilot study examining the effects of exercise on mood, learning, memory, attention, stress, and sleeping habits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Running group (Experimental): 13 week, bi-weekly running group
  Interventions: Other: Running

INTERVENTIONS:
Other: Running — A 13-week running program where youth run for 30 minutes twice weekly.
  Other Names: Exercise

SUMMARY:
The investigators are interested in finding accessible interventions for youth and young adults that help promote long-term positive mental health functioning. They will be investigating the effects of Team Unbreakable, a 13-week, twice weekly running group, on mental health symptoms, memory, and attention. This intervention will hopefully improve mental health functioning in youth aged 17-25 that are at high risk of developing mental health disorders. Sessions will consist of 30 minutes of running under the supervision of group leaders and coaches. The group will steadily increase the distance and time spent running versus walking, with the goal of having everyone run a 5 km race together at the end of 13 weeks. Once a week, youth will be provided with education on a variety of topics related to health and running. Youth will complete measures before, during, and after the program to assess outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy enough to participate in physical activity

Exclusion Criteria:

* NOT excluded on basis of mental health or addiction concerns

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ-9) | Starting 1 month to 2 weeks prior to group. Administered on a bi-weekly schedule ending 6 months after the conclusion of the running group.
  Nine-item self-report measure designed to monitor the severity of depressive symptoms using the diagnostic criteria found in the DSM-IV
Generalized Anxiety Disorder 7 (GAD-7) | Starting 1 month to 2 weeks prior to group. Administered on a bi-weekly schedule ending 6 months after the conclusion of the running group.
  Seven-item self-report anxiety questionnaire designed to monitor and assess the severity of generalized anxiety disorder (GAD) symptoms, using the prominent diagnostic features found in the DSM-IV
Kessler Psychological Distress Scale (K-10) | Starting 1 month to 2 weeks prior to group. Administered on a 4-week schedule ending 6 months after the conclusion of the running group.
  Ten-item self-report measure of global psychological distress

SECONDARY OUTCOMES:
PTSD Checklist for DSM-V (PCL-5) | Starting 1 month to 2 weeks prior to group. Administered on a 4-week schedule ending 6 months after the conclusion of the running group.
  Twenty-item self-report measure of PTSD based on the DSM-V diagnostic criteria
Rosenberg Self-Esteem Scale (RSES) | Starting 1 month to 2 weeks prior to group. Administered on a 4-week schedule ending 6 months after the conclusion of the running group.
  Ten-item self-report measure of global feelings of self-worth
Multidimensional Scale of Perceived Social Support | Starting 1 month to 2 weeks prior to group. Administered on a 4-week schedule ending 6 months after the conclusion of the running group.
  Twelve-item self-report measure of perceived support from three sources: Family, friends, and a significant other
Work and Social Adjustment Scale (WSAS) | Starting 1 month to 2 weeks prior to group. Administered on a 4-week schedule ending 6 months after the conclusion of the running group.
  Five-item self-report measure of impairment in functioning
Physical Activity and Sleep | Starting 1 month to 2 weeks prior to group auto-recorded ending 6 months after the conclusion of the running group.
  Participants will use a Fitbit to monitor their overall activity (e.g., steps, distance, active minutes, etc.) and sleep patterns before, during, and after treatment
Delis-Kramer Executive Function Tower Task | At baseline and 1-week after exercise program ends.
  Assesses spatial planning, rule learning, and response inhibition
Hopkins Verbal Learning Task | At baseline and 1-week after exercise program ends.
  Tests participants' memory for a list of 12 nouns drawn from 3 categories, and measures immediate and delayed recall and recognition
N-back | At baseline and 1-week after exercise program ends.
  A test of executive function (working memory), requiring the participant to observe a sequence of items and click on targets that are repeats n items ago
Concentration Memory Task | At baseline and 1-week after running program ends.
  A test of high interference spatial memory. Participants search for pairs of matching cards and are periodically tested on which of two locations an item appeared in most recently
Town Square | At baseline and 1-week after running program ends.
  A test of viewpoint-dependent and -independent spatial memory for a set of visually presented items in a town square
Wechsler Test of Adult Reading | At baseline
  A test to assess pre-morbid intellectual functioning by having the participants verbally speak a list of 50 irregular words

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Tobon, PhD, CPsych, Principal Investigator — St. Joseph's Research Institute - Youth Wellness Centre
Locations (1):
- Youth Wellness Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] RiskAnalytica. The life and economic impact of major mental illnesses in canada. Mental Health Commission of Canada. 2011:2011-2041.
- [Background] Lim KL, Jacobs P, Ohinmaa A, Schopflocher D, Dewa CS. A new population-based measure of the economic burden of mental illness in Canada. Chronic Dis Can. 2008;28(3):92-8. PMID 18341763
- [Background] Merikangas KR, Nakamura EF, Kessler RC. Epidemiology of mental disorders in children and adolescents. Dialogues Clin Neurosci. 2009;11(1):7-20. doi: 10.31887/DCNS.2009.11.1/krmerikangas. PMID 19432384
- [Background] Shapiro CM, Bortz R, Mitchell D, Bartel P, Jooste P. Slow-wave sleep: a recovery period after exercise. Science. 1981 Dec 11;214(4526):1253-4. doi: 10.1126/science.7302594.
- [Background] Dery N, Pilgrim M, Gibala M, Gillen J, Wojtowicz JM, Macqueen G, Becker S. Adult hippocampal neurogenesis reduces memory interference in humans: opposing effects of aerobic exercise and depression. Front Neurosci. 2013 Apr 30;7:66. doi: 10.3389/fnins.2013.00066. eCollection 2013. PMID 23641193
- [Background] Anderson RJ, Brice S. The mood-enhancing benefits of exercise: Memory biases augment the effect. Psychology of Sport & Exercise. 2011;12(2):79-82. doi: 10.1016/j.psychsport.2010.08.003.
- [Background] van Oers HM. Exercise effects on mood in breast cancer patients. South African Journal of Sports Medicine. 2013;25(2):55. doi: 10.7196/SAJSM.481.
- [Background] Prakash RS, Voss MW, Erickson KI, Lewis JM, Chaddock L, Malkowski E, Alves H, Kim J, Szabo A, White SM, Wojcicki TR, Klamm EL, McAuley E, Kramer AF. Cardiorespiratory fitness and attentional control in the aging brain. Front Hum Neurosci. 2011 Jan 14;4:229. doi: 10.3389/fnhum.2010.00229. eCollection 2011. PMID 21267428
- [Background] Chang YK, Pesce C, Chiang YT, Kuo CY, Fong DY. Antecedent acute cycling exercise affects attention control: an ERP study using attention network test. Front Hum Neurosci. 2015 Apr 9;9:156. doi: 10.3389/fnhum.2015.00156. eCollection 2015. PMID 25914634
- [Background] Monti JM, Hillman CH, Cohen NJ. Aerobic fitness enhances relational memory in preadolescent children: the FITKids randomized control trial. Hippocampus. 2012 Sep;22(9):1876-82. doi: 10.1002/hipo.22023. Epub 2012 Apr 23. PMID 22522428
- [Background] Quelhas Martins A, Kavussanu M, Willoughby A, Ring C. Moderate intensity exercise facilitates working memory. Psychology of Sport and Exercise. 2013;14(3):323-328. doi: 10.1016/j.psychsport.2012.11.010
- [Background] Guiney H, Machado L. Benefits of regular aerobic exercise for executive functioning in healthy populations. Psychon Bull Rev. 2013 Feb;20(1):73-86. doi: 10.3758/s13423-012-0345-4. PMID 23229442
- [Background] Snyder JS, Soumier A, Brewer M, Pickel J, Cameron HA. Adult hippocampal neurogenesis buffers stress responses and depressive behaviour. Nature. 2011 Aug 3;476(7361):458-61. doi: 10.1038/nature10287. PMID 21814201
- [Background] van Praag H, Shubert T, Zhao C, Gage FH. Exercise enhances learning and hippocampal neurogenesis in aged mice. J Neurosci. 2005 Sep 21;25(38):8680-5. doi: 10.1523/JNEUROSCI.1731-05.2005. PMID 16177036
- [Background] Hutton CP, Dery N, Rosa E, Lemon JA, Rollo CD, Boreham DR, Fahnestock M, deCatanzaro D, Wojtowicz JM, Becker S. Synergistic effects of diet and exercise on hippocampal function in chronically stressed mice. Neuroscience. 2015 Nov 12;308:180-93. doi: 10.1016/j.neuroscience.2015.09.005. Epub 2015 Sep 7. PMID 26358368
- [Background] Nuechterlein KH, Dawson ME, Ventura J, Gitlin M, Subotnik KL, Snyder KS, Mintz J, Bartzokis G. The vulnerability/stress model of schizophrenic relapse: a longitudinal study. Acta Psychiatr Scand Suppl. 1994;382:58-64. doi: 10.1111/j.1600-0447.1994.tb05867.x. PMID 8091999
- [Background] Alexander SJ, Harrison AG. Cognitive responses to stress, depression, and anxiety and their relationship to ADHD symptoms in first year psychology students. J Atten Disord. 2013 Jan;17(1):29-37. doi: 10.1177/1087054711413071. Epub 2011 Aug 8. PMID 21825110
- [Background] Sinha R. Modeling stress and drug craving in the laboratory: implications for addiction treatment development. Addict Biol. 2009 Jan;14(1):84-98. doi: 10.1111/j.1369-1600.2008.00134.x. Epub 2008 Oct 20. PMID 18945295
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Gilbody S, Richards D, Brealey S, Hewitt C. Screening for depression in medical settings with the Patient Health Questionnaire (PHQ): a diagnostic meta-analysis. J Gen Intern Med. 2007 Nov;22(11):1596-602. doi: 10.1007/s11606-007-0333-y. Epub 2007 Sep 14. PMID 17874169
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Kessler RC, Andrews G, Colpe LJ, Hiripi E, Mroczek DK, Normand SL, Walters EE, Zaslavsky AM. Short screening scales to monitor population prevalences and trends in non-specific psychological distress. Psychol Med. 2002 Aug;32(6):959-76. doi: 10.1017/s0033291702006074. PMID 12214795
- [Background] Dal Grande E, Taylor A, Wilson D. South australian health and wellbeing survey, december 2000. Centre for Population Studies in Epidemiology. 2002.
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Rosenberg M. Society and the adolescent self-image. Princeton, NJ: Univ. Press; 1965.
- [Background] Bagley C, Bolitho F, Bertrand L. Norms and construct validity of the rosenberg self-esteem scale in canadian high school populations: Implications for counselling. Canadian Journal of Counselling. 1997;31(1):82.
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Canty-Mitchell J, Zimet GD. Psychometric properties of the Multidimensional Scale of Perceived Social Support in urban adolescents. Am J Community Psychol. 2000 Jun;28(3):391-400. doi: 10.1023/A:1005109522457. PMID 10945123
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Michael E. Sobel. Asymptotic confidence intervals for indirect effects in structural equation models. Sociological Methodology. 1982;13:290-312.
- See also: Mental and substance use disorders in canada. — http://www.statcan.gc.ca/pub/82-624-x/2013001/article/11855-eng.htm
- See also: Greenspace Mental Health Ltd. — https://www.grnspace.com/
- See also: PTSD checklist for DSM-5 (PCL-5) made available from the National Center for PTSD. — http://www.ptsd.va.gov